CLINICAL TRIAL: NCT07350096
Title: The Effects of Intensive Physiotherapy on Postural Control and Selective Motor Control of the Upper and Lower Extremities in Children With Spastic Cerebral Palsy
Brief Title: The Effects of Intensive Physiotherapy in Children With Spastic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Fatma Hazal Ağbaba, Clinical Physiotherapist, MSc. Physiotherapist, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10840098-604.01.01-E.5016
Record Dates: First submitted 2025-12-28; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Cerebral Palsy (CP)
Keywords: cerebral palsy; intensive therapy; selective motor control; postural control; neurodevelopmental treatment
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Physiotherapy Program (Experimental): Participants in the experimental group received a 2-week intensive physiotherapy program based on Neurodevelopmental Treatment (NDT) principles with active participation.
  Frequency: 6 days per week Sessions: 2 sessions per day Session duration: 50 minutes Total sessions: 24
  Intervention components included:
  * Weight-shifting and reaching activities in crawling, sitting, kneeling, and standing positions
  * Functional and symmetrical reaching tasks in different postures
  * Actively assisted transitions between postures
  * Balance training and facilitation of protective reactions in various positions
  * Core stabilization exercises
  * Isolated strengthening exercises for upper and lower extremities
  * Proprioceptive training exercises
  Interventions: Behavioral: Neurodevelopmental Therapy
- Conventional Physiotherapy Program (Experimental): Participants in the control group received a 2-week conventional physiotherapy program.
  Frequency: 3 days per week Sessions: 1 session per day Session duration: 45 minutes Total sessions: 6
  Intervention components included:
  * Stretching and strengthening exercises
  * Passive and active range of motion exercises
  * Balance and coordination exercises in different positions
  * Electrotherapy applications
  Interventions: Behavioral: Conventional Therapy

INTERVENTIONS:
Behavioral: Neurodevelopmental Therapy — Intervention components included:
  * Weight-shifting and reaching activities in crawling, sitting, kneeling, and standing positions
  * Functional and symmetrical reaching tasks in different postures
  * Actively assisted transitions between postures
  * Balance training and facilitation of protective reactions in various positions
  * Core stabilization exercises
  * Isolated strengthening exercises for upper and lower extremities
  * Proprioceptive training exercises
  Frequency: 6 days per week Sessions: 2 sessions per day Session duration: 50 minutes Total sessions: 24
  Arms: Intensive Physiotherapy Program
Behavioral: Conventional Therapy — Intervention components included:
  * Stretching and strengthening exercises
  * Passive and active range of motion exercises
  * Balance and coordination exercises in different positions
  * Electrotherapy applications
  Frequency: 3 days per week Sessions: 1 session per day Session duration: 45 minutes Total sessions: 6
  Arms: Conventional Physiotherapy Program

SUMMARY:
The aim of this study is to investigate the effects of a 2-week Neurodevelopmental Treatment (NDT)-based intensive physiotherapy program with active participation on postural control and selective motor control of the lower and upper extremities in children diagnosed with spastic cerebral palsy.

Thirty children with spastic type cerebral palsy, aged between 4 and 8 years, and classified as level II, III, or IV according to the Gross Motor Function Classification System (GMFCS), will be included in the study. Participants will be randomized into two groups.

The experimental group will receive an NDT-based intensive physiotherapy program with active participation for 2 weeks, 6 days per week, 2 sessions per day, with each session lasting 50 minutes. The control group will receive a conventional physiotherapy program for 2 weeks, 3 days per week, once per day, with each session lasting 45 minutes.

Outcome measures will be assessed before and after the intervention period and will include the Seated Postural Control Measure-Function (SPCM-Function), Selective Control Assessment of the Lower Extremity (SCALE), Selective Control of the Upper Extremity Scale (SCUES), Modified Ashworth Scale (MAS), Gross Motor Function Measure-88 (GMFM-88) and the Pediatric Quality of Life Inventory (PedsQL).

DETAILED DESCRIPTION:
This study was not prospectively registered in a public trials registry. Registration was completed retrospectively after data collection had been completed.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4-8 years,
* No Botulinum Toxin type A injections within the last 6 months,
* No orthopedic surgical intervention within the last 12 months,
* Able to understand simple verbal commands and cooperate,
* Diagnosed with cerebral palsy,
* Spastic clinical type,
* Classified as Gross Motor Function Classification System (GMFCS) levels II, III, and IV.

Exclusion Criteria:

* Failure to participate regularly in the treatment program,
* Failure to participate in pre- and post-treatment assessments,
* Children who were severely distressed, crying excessively, or uncooperative.
* Children who have cognitive problems,
* Children who have active seizures.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Seated Postural Control Measure | Baseline (pre-intervention) and immediately after completion of the 2-week intervention.
  Seated Postural Control Measure (SPCM) evaluates static, active, and reactive trunk control at different trunk segments in a supported sitting position. It identifies the highest trunk level at which independent postural control is achieved in children with cerebral palsy. SPCM consists of three sub scales. In this study only function subscale will be used. The Function subscale of the Seated Postural Control Measure consists of 12 items evaluating head and trunk control during sitting, reaching, grasping and releasing, bimanual use, and wheelchair mobility. Each item is scored on a 4-point ordinal scale ranging from 1 to 4 points, with higher scores indicating better task performance. The total score of the Function subscale ranges from a minimum of 12 points to a maximum of 48 points.
The Selective Motor Control of the Upper Extremity | Baseline (pre-intervention) and immediately after completion of the 2-week intervention.
  The Selective Control of the Upper Extremity Scale (SCUES) selective voluntary motor control of the shoulder, elbow, forearm, wrist, and fingers during functional tasks in children with cerebral palsy. Higher scores indicate better selective motor control of the upper extremities.Selective motor control (SMC) is graded for each joint using a four-point ordinal scale: 3 points indicate normal selective motor control, 2 points- mildly impaired SMC, 1 point-moderately impaired SMC, 0 points- absence of SMC. For each upper extremity maximum point is 15.
The Selective Motor Control of the Lower Extremity | Baseline (pre-intervention) and immediately after completion of the 2-week intervention.
  The Selective Control Assessment of the Lower Extremity (SCALE) evaluates the ability to perform isolated voluntary movements at the hip, knee, ankle, subtalar joint, and toes independently of mass synergistic patterns in children with cerebral palsy.Higher scores indicate better SMC of the lower extremities.2 points- normal SMC, 1point impaired SMC, and 0 points unable to perform. For each lower extremity maximum point is 10.

SECONDARY OUTCOMES:
Gross Motor Function Measure-88 (GMFM-88) | Baseline (pre-intervention) and immediately after completion of the 2-week intervention.
  The Gross Motor Function Measure-88 (GMFM-88) evaluates changes in gross motor function, including lying and rolling, sitting, crawling and kneeling, standing, and walking, running, and jumping in children with cerebral palsy. The Gross Motor Function Measure-88 consists of 88 items and is administered through observation of motor performance by a physiotherapist in children with cerebral palsy.
  Each item is scored on a 4-point ordinal scale as follows:
  0 - Does not initiate the movement,
  1. - Initiates the movement (<10% of the task),
  2. - Partially completes the movement (10-90% of the task),
  3. - Completes the movement independently. Scores for each dimension are calculated as percentages. The total GMFM-88 score is obtained by averaging the five dimension percentage scores (0-100). Higher percentage scores indicate better gross motor function.
Modified Ashworth Scale (MAS) | Baseline (pre-intervention) and immediately after completion of the 2-week intervention.
  The Modified Ashworth Scale (MAS) assesses muscle spasticity of the upper and lower extremities by measuring resistance during passive movement. Muscle tone is assessed using the Modified Ashworth Scale, which grades resistance to passive movement on an ordinal scale ranging from 0 to 4, where 0 indicates no increase in muscle tone and 4 indicates rigidity in flexion and extension of the affected part. Higher scores indicating greater spasticity.
Pediatric Quality of Life Inventory (PedsQL) | Baseline (pre-intervention) and immediately after completion of the 2-week intervention.
  The Pediatric Quality of Life Inventory assesses health-related quality of life in children with cerebral palsy through age-appropriate parent-report and child self-report forms.Items on the Pediatric Quality of Life Inventory (PedsQL) Generic Core Scales are reverse scored and linearly transformed to a 0-100 scale, where higher scores indicate better health-related quality of life. Item scoring is performed as follows:
  0 ("Never") = 100
  1. ("Almost Never") = 75
  2. ("Sometimes") = 50
  3. ("Often") = 25
  4. ("Almost Always") = 0 Scale scores are calculated as the mean of the completed item scores. To account for missing data, a scale score is computed only if at least 50% of the items are completed. If more than 50% of items are missing, the scale score is not calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Department of Physiotherapy and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wimalasundera N, Stevenson VL. Cerebral palsy. Pract Neurol. 2016 Jun;16(3):184-94. doi: 10.1136/practneurol-2015-001184. Epub 2016 Feb 2. PMID 26837375
- [Result] Fowler EG, Staudt LA, Greenberg MB, Oppenheim WL. Selective Control Assessment of the Lower Extremity (SCALE): development, validation, and interrater reliability of a clinical tool for patients with cerebral palsy. Dev Med Child Neurol. 2009 Aug;51(8):607-14. doi: 10.1111/j.1469-8749.2008.03186.x. Epub 2009 Feb 12. PMID 19220390
- [Result] Palisano RJ, Rosenbaum P, Bartlett D, Livingston MH. Content validity of the expanded and revised Gross Motor Function Classification System. Dev Med Child Neurol. 2008 Oct;50(10):744-50. doi: 10.1111/j.1469-8749.2008.03089.x. PMID 18834387
- [Result] Choi JY. Motor Function Measurement in Children: Gross Motor Function Measure (GMFM). Ann Rehabil Med. 2024 Oct;48(5):301-304. doi: 10.5535/arm.240078. Epub 2024 Oct 2. No abstract available. PMID 39354669
- [Result] Mutlu A, Livanelioglu A, Gunel MK. Reliability of Ashworth and Modified Ashworth scales in children with spastic cerebral palsy. BMC Musculoskelet Disord. 2008 Apr 10;9:44. doi: 10.1186/1471-2474-9-44. PMID 18402701
- [Result] Wagner LV, Davids JR, Hardin JW. Selective Control of the Upper Extremity Scale: validation of a clinical assessment tool for children with hemiplegic cerebral palsy. Dev Med Child Neurol. 2016 Jun;58(6):612-7. doi: 10.1111/dmcn.12949. Epub 2015 Nov 3. PMID 26526592
- [Result] Varni JW, Burwinkle TM, Berrin SJ, Sherman SA, Artavia K, Malcarne VL, Chambers HG. The PedsQL in pediatric cerebral palsy: reliability, validity, and sensitivity of the Generic Core Scales and Cerebral Palsy Module. Dev Med Child Neurol. 2006 Jun;48(6):442-9. doi: 10.1017/S001216220600096X. PMID 16700934
- [Result] Gulati S, Sondhi V. Cerebral Palsy: An Overview. Indian J Pediatr. 2018 Nov;85(11):1006-1016. doi: 10.1007/s12098-017-2475-1. Epub 2017 Nov 20. PMID 29152685
- [Result] Santamaria V, Rachwani J, Saussez G, Bleyenheuft Y, Dutkowsky J, Gordon AM, Woollacott MH. The Seated Postural & Reaching Control Test in Cerebral Palsy: A Validation Study. Phys Occup Ther Pediatr. 2020;40(4):441-469. doi: 10.1080/01942638.2019.1705456. Epub 2020 Jan 3. PMID 31900006
- [Result] Balzer J, van der Linden ML, Mercer TH, van Hedel HJA. Selective voluntary motor control measures of the lower extremity in children with upper motor neuron lesions: a systematic review. Dev Med Child Neurol. 2017 Jul;59(7):699-705. doi: 10.1111/dmcn.13417. Epub 2017 Mar 8. PMID 28272744
- [Result] Hong BY, Jo L, Kim JS, Lim SH, Bae JM. Factors Influencing the Gross Motor Outcome of Intensive Therapy in Children with Cerebral Palsy and Developmental Delay. J Korean Med Sci. 2017 May;32(5):873-879. doi: 10.3346/jkms.2017.32.5.873. PMID 28378564
- [Result] Lee H, Kim EK, Son DB, Hwang Y, Kim JS, Lim SH, Sul B, Hong BY. The Role of Regular Physical Therapy on Spasticity in Children With Cerebral Palsy. Ann Rehabil Med. 2019 Jun;43(3):289-296. doi: 10.5535/arm.2019.43.3.289. Epub 2019 Jun 28. PMID 31311250
- [Result] Park EY. Path analysis of strength, spasticity, gross motor function, and health-related quality of life in children with spastic cerebral palsy. Health Qual Life Outcomes. 2018 Apr 19;16(1):70. doi: 10.1186/s12955-018-0891-1. PMID 29673348
- [Result] Sukal-Moulton T, Gaebler-Spira D, Krosschell KJ. The validity and reliability of the Test of Arm Selective Control for children with cerebral palsy: a prospective cross-sectional study. Dev Med Child Neurol. 2018 Apr;60(4):374-381. doi: 10.1111/dmcn.13671. Epub 2018 Jan 31. PMID 29383702
- [Result] Tuncdemir M, Unes S, Karakaya J, Kerem Gunel M. Reliability and validity of the Turkish version of the Selective Control Assessment of the Lower Extremity (SCALE) in children with spastic cerebral palsy. Disabil Rehabil. 2023 Jan;45(1):106-110. doi: 10.1080/09638288.2021.2022783. Epub 2022 Jan 7. PMID 34994671